CLINICAL TRIAL: NCT01967693
Title: Characterization of Laryngeal Contact Granulomas: Retrospective Analysis of Symptoms, Promotive Factors and Therapy
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BJ_04_04_2012
Record Dates: First submitted 2013-09-18; First posted 2013-10-23 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Laryngeal Contact Granuloma
Keywords: Laryngeal contact granuloma; Treatment type; Outcome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Retrospective analysis of data — Retrospective data analysis

SUMMARY:
Retrospective analysis of data from patients with laryngeal contact granulomas in order to identify possible differences and/or similarities between the cases and in order to determine whether and which conclusions can be drawn on disease and therapy.

DETAILED DESCRIPTION:
This is a retrospective analysis of data from patients with laryngeal contact granulomas in order to identify possible differences and/or similarities between the cases and in order to determine whether and which conclusions can be drawn on disease and therapy.

ELIGIBILITY:
Inclusion criteria:

Laryngeal contact granuloma in adults with documentation of symptoms, possible causes, therapy and outcome

Exclusion criteria:

Incomplete information on the diagnosis laryngeal contact granuloma (symptoms, promotive factors, findings)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former patients with laryngeal contact granuloma who were treated in this hospital.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with similar therapy outcome as a measure of therapy predictability | 4 to 6 months after finishing the therapy
  Data from patients with laryngeal contact granuloma are analyzed retrospectively as to wether similar pathologies and treatment lead to similar outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg E. Bohlender, KD Dr. med., Principal Investigator — University Hospital Zurich, Division of Otorhinolaryngology
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology, Zurich, Canton of Zurich, Switzerland